CLINICAL TRIAL: NCT05434832
Title: The Effect of Virtual Reality and Local Cold Application-Vibration Methods on Reducing Anxiety, Fear and Pain Developed During Intramuscular Injection in Children
Brief Title: Effects of Virtual Reality, External Cold and Vibration to Children During IM Injection on Pain, Fear and Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ozge Denli Ozgen, Nurse, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019/920; 5207 (Other Grant/Funding Number: AKD Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2022-06-16; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Procedural Pain; Fear; Procedural Anxiety; Child, Only
Keywords: child; pain; anxiety; fear; intramuscular injection; local cold-vibration; virtual reality; pediatric nurse
MeSH Terms: conditions — Pain, Procedural; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A total of three groups as 2 intervention (virtual reality, local cold-vibration) and control group (routine application)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Group (Experimental): watching the cartoon by wearing virtual reality glass to the child during the intramuscular injection
  Interventions: Behavioral: Virtual Reality
- Local cold-vibration Group (Experimental): The local cold-vibration device is placed 5 cm above the area to be injected
  Interventions: Behavioral: Local cold-vibration
- Control Group (No Intervention): standart care

INTERVENTIONS:
Behavioral: Virtual Reality — Distraction method
  Arms: Virtual Reality Group
Behavioral: Local cold-vibration — Distraction method
  Arms: Local cold-vibration Group

SUMMARY:
A randomized controlled trial is conducted to evaluation of the effects of virtual reality and local cold-vibration applications in reducing anxiety, fear and pain due to intramuscular (IM) injection in children aged 5-10 years. It has been determined that the use of Virtual Reality and local cold-vibration are effective interventions in reducing anxiety, fear and pain due to IM injection in children aged 5-10 years.

DETAILED DESCRIPTION:
Intramuscular (IM) intervention is a parenteral administration method that is frequently used in children and causes pain. In cases such as inadequacies in pain management and inability to prevent pain, physiological and psychological problems that can last a lifetime can be seen in the child. There are different non-pharmacological methods for reducing pain due to invasive procedures. The use of non-pharmacological methods is an important part of nursing care to reduce the short and long-term negative effects of painful interventions on children. However, the use of non-pharmacological methods to reduce the pain perceived by the child during painful interventions in pediatric emergency units is not common in our country. No study has been found in the literature comparing the effectiveness of virtual reality and Buzzy methods in reducing anxiety, fear and pain due to invasive procedures. This study was planned to compare the effectiveness of virtual reality and local cold application-vibration applications in reducing anxiety, fear and pain caused by intramuscular injection in children aged 5-10 years. It was planned as a randomized controlled experimental study in pre-test, post-test design. The sample of the study was carried out in the Pediatric Emergency Unit of Konya Selcuk University Medical Faculty Hospital. The applicant will consist of 120 children aged 5-10 years. There will be a total of three groups in the research, 2 of which are the intervention group (virtual reality, Buzzy) and the control group (routine application). Data will be collected using the "Child-Parent Description Form", "Child Anxiety Scale-State Scale", "Child Fear Scale", "Wong- Baker Faces Pain Scale". Data will be collected before and within the first 5 minutes after IM injection administration. Scales; to be filled in separately by the child, one of the parents, and the nurse administering the IM injection. As a result of this study, it was concluded that the use of virtual reality glasses and local cold application-vibration (Buzzy) methods are effective in reducing the pain, anxiety and fear that develop during IM injection in children aged 5-10 years.

ELIGIBILITY:
Inclusion Criteria:

The child is between the ages of 5 and 10

Having intramuscular (IM) injection therapy

Absence of Audio-Visual-Sensation loss problem

No communication problem

Absence of mental retardation

Absence of a disease causing chronic pain

No history of fainting during injection

Not taking any analgesic medication in the last 4 hours

Exclusion Criteria:

Failure of IM application at one time

The child in the virtual reality application group removes the virtual reality glasses during the IM injection.

The child in the group receiving Buzzy application removes the Buzzy device during IM injection.

Not wanting to fill the scales after the application

Diagnosis or suspicion of COVID-19 (having any of the symptoms such as fever, cough, respiratory distress, chest pain, loss of taste and smell, sore throat, contact with a COVID-19 positive person)

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-06-27 (Estimated)

PRIMARY OUTCOMES:
Anxiety assesed by Children's State Anxiety | Before the intramuscular injection
  The Children's State Anxiety (CAS-S). The CAS-S assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety
Anxiety assesed by Children's State Anxiety | Within the first 5 minutes after the intramuscular injection
  The Children's State Anxiety (CAS-S). The CAS-S assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety
Fear assesed by Child Fear Scale | Before the intramuscular injection
  The Child Fear Scale (CFS). The Child Fear Scale will use.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear. This rating scale ranges from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome. The rater responds indicates the level of fear.
Fear assesed by Child Fear Scale | Within the first 5 minutes after the intramuscular injection
  The Child Fear Scale (CFS). The Child Fear Scale will use.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear. This rating scale ranges from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome. The rater responds indicates the level of fear.
Pain assesed by Wong-Baker FACES | Before the intramuscular injection
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Pain assesed by Wong-Baker FACES | Within the first 5 minutes after the intramuscular injection
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).

CONTACTS AND LOCATIONS:
Overall Officials: AYŞEGÜL İŞLER DALGIÇ, Professor, Study Director — Akdeniz University
Locations (1):
- Ayşegül İşler Dalgiç, Antalya, Akdeniz University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No